CLINICAL TRIAL: NCT02183181
Title: A Randomized, Single-dose, Two-way Crossover Study to Assess the Bioequivalence of Meloxicam Capsules 15 mg (Mobic® Capsules 15 mg) Versus Meloxicam Tablets 15 mg (Mobic® Tablets 15 mg) Administered to Healthy Adult Volunteers
Brief Title: Bioequivalence Study of Meloxicam Capsules 15 mg (Mobic® Capsules 15 mg) Versus Meloxicam Tablets 15 mg (Mobic® Tablets 15 mg) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.274
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

ARMS (2):
- Meloxicam capsule (Experimental): Capsules 15 mg
  Interventions: Drug: Meloxicam capsule
- Meloxicam tablet (Active Comparator): Tablets 15 mg
  Interventions: Drug: Meloxicam tablet

INTERVENTIONS:
Drug: Meloxicam capsule
  Arms: Meloxicam capsule
Drug: Meloxicam tablet
  Arms: Meloxicam tablet

SUMMARY:
Primary Objective:

To access the bioequivalence of meloxicam capsule 15 mg (Test, T) to meloxicam tablet 15mg (Reference, R) following oral administration.

Secondary Objective:

To investigate the safety and tolerability of meloxicam following a single dose of meloxicam capsule 15 mg vs. meloxicam tablet 15 mg under fasting conditions in healthy male Taiwanese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent before enrolment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study
2. Healthy adult male, aged between 20 and 40 years old
3. Body Mass Index (BMI) between 18.5 and 25, inclusive (BMI was calculated as weight in kilogram [kg]/height in meters2 [m2]).
4. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest x-ray and electrocardiogram.
5. No significant deviation from biochemistry including: aspartate transaminase (SGOT/AST), alanine transaminase (SGPT/ALT), gamma-glutamyl-transferase (GGT), alkaline phosphatase, total bilirubin, albumin, glucose, blood urea nitrogen (BUN), creatinine, uric acid, total cholesterol and triglyceride.
6. No significant deviation from normal hematology including: hemoglobin, hematocrit, white blood count (WBC) with differential, red blood count (RBC) and platelet count
7. No significant deviation from normal urinalysis including: pH, occult blood, glucose and protein.

Exclusion Criteria:

1. History of drug or alcohol abuse within the past one year
2. Medical history of allergic asthma or sensitivity to analogous drug
3. Evidence of chronic or acute infectious diseases from 4 weeks before the study
4. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology.
5. Ongoing peptic ulcer and constipation
6. Planned vaccination during the time course of the study.
7. Taking any clinical investigation drug from 3 months before the study
8. Use of any medication, including herb medicine or vitamins from 4 weeks before the study
9. Blood donation of more than 500 ml within the past 3 months
10. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result
11. A positive test for HIV antibody

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval zero to infinity (AUC0-infinity) | 0, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24, 48, 72 and 96 hours after administration
Area under the plasma concentration-time curve from 0 h to last concentration time (AUC0-tz) | 0, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24, 48, 72 and 96 hours after administration
Observed maximum measured concentration of the analyte in plasma (Cmax) | 0, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24, 48, 72 and 96 hours after administration
Time to reach maximum plasma concentration (Tmax) | 0, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24, 48, 72 and 96 hours after administration
Plasma half-life estimated by (0.693/ kel) ( t ½) | 0, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24, 48, 72 and 96 hours after administration

SECONDARY OUTCOMES:
Occurrence of adverse events | up to 33 days after first administration
Drug induced changes in standard laboratory values | screening phase (at least 10hours fasting), before and 24 h following drug administration on each study day, within 14 days after completion of all two periods